CLINICAL TRIAL: NCT04519606
Title: Optimization of Respiratory Mechanics During One-lung Ventilation
Brief Title: Respiratory Mechanics During One-lung Ventilation
Status: Completed | Type: Observational
Sponsor: E-DA Hospital (Other)
Responsible Party: Principal Investigator, Tu, Yuan-Kun, Superintendent, professor, E-DA Hospital
Other Study IDs: EMRP69108N
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Ventilator-Induced Lung Injury; Lung Ventilator; One-lung Ventilation
Keywords: Barotrauma; Volutrauma; Biotrauma; Atelectasis; Lung recruitment
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Barotrauma; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One-lung ventilation: During one-lung ventilation, the dependent lung (non-operation lung) will be mechanically ventilated with a fixed positive end-expiratory pressure (PEEP) of 4 cmH2O and the peak pressure below 30 cmH2O. Tidal volumes will be titrated from the initial 4 ml/kg predicted body weight (PBW) to 7 ml/kg PBW. Optimal lung compliance is determined by the levels of upper reflection point of the pressure-volume loop closed to 30 cmH2O. Chest tomography will be undertaken with the optimal tidal volume during OLV phase and when the independent lung is completely recruited using the stepwise PEEP increase method.
  Interventions: Procedure: Optimal lung compliance during OLV

INTERVENTIONS:
Procedure: Optimal lung compliance during OLV — Stepwise increase of tidal volume from 4 ml/kg PBW to 7 ml/kg PBW during OLV to determine the optimal tidal volume at the level the the pressure-volume loop reaches upper refection point where the peak airway pressure at or just below 30 cmH2O

SUMMARY:
Intraoperative lung protective ventilatory strategy has been widely recognized to reduce postoperative pulmonary complications in laparotomy and laparoscopic surgeries. However, the clinical evidence and consensus for ventilatory strategy to protect the dependent lung segments during thoracic surgery that requires one-lung ventilation (OLV) is currently not available. Since lung compliance changes significantly during OLV, the levels of respiratory mechanics should be optimized to avoid barotrauma and volutrauma. This study aims to determine the optimal levels of volume-pressure dynamics during OLV and at the phase of recruitment of the independent lungs by achieving optimal lung compliance, gas exchange and hemodynamics.

DETAILED DESCRIPTION:
Background One-lung ventilation (OLV) is the foremost used technique of ventilation during thoracic procedures. Intraoperative lung separation can be managed by means of double-lumen endotracheal tube (DLT), bronchial blocker (BB), or nonintubated method. OLV is impeded by significant reduction in lung volume, decline in lung compliance at lateral decubital position, formation of intrapulmonary shunting and exposure of the dependent lung to ventilator-induced lung injury (VILI). In addition, patients receiving thoracic surgeries are more prone to developing acute lung injuries due to direct surgery-related trauma caused by instrumentation or manipulation of the lung tissues, hypoperfusion induced by hypoxic pulmonary vasoconstriction, and dysfunction of surfactant system. The non-dependent lung is injured by surgical manipulation and atelectrauma. Re-expansion of the collapsed non-dependent lung at the end of surgery inevitably results in systemic inflammatory response in the local and contralateral lungs, which in turn leads to biotrauma. Therefore, a significantly high pulmonary complication of up to 14-28.4% was reported in patients that received OLV surgery.

In the recent two decades, there is a major paradigm shift for mechanical ventilator support during operation by the introduction of intraoperative lung protective ventilation strategies. Some of these changes include a low tidal volume (Vt), moderate levels of positive end-expiratory pressure (PEEP), optimal driving pressure (∆P) and the appropriate use of lung recruitment maneuver. Intraoperative lung protective ventilation strategies have been shown to reduce post-operative pulmonary complications and improve overall clinical outcomes in intermediate and high-risk patients undergoing major abdominal surgery. Currently, however, there is a lack of clinical evidence in regard to appropriate protective-lung strategies during OLV. The optimal levels of intraoperative use of oxygen fraction, the ventilatory settings for volume and pressure variables during OLV and re-expansion phases for lung recruitment are debating. The main objective of this clinical study is to determine the optimal levels of volume-pressure dynamics during OLV and at the phase of recruitment of the independent lungs by achieving optimal lung compliance, gas exchange and hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for single lobectomy or wedge resection of right or left lung lobe
* American Society of Anesthesiologists physical classification (ASA PC) I-III
* Preoperative normal pulmonary function test

Exclusion Criteria:

* Anticipated difficult intubation or ventilation
* Severe heart failure (NYHA Fc >=3)
* Advanced liver cirrhosis (Child-Pugh score >=B)
* Advanced renal disease (creatinine >2 mg/dl)
* Severe anemia (hemoglobin <8 mg/dl)
* Body mass index >30
* Pregnancy
* Emergency operation
* Prior history of heart, lung or mediastinal surgery
* Psychiatric or other mental disorders
* Patient refusal

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Generally healthy (ASA PC I-III) patients receiving thoracic surgery that required intraoperative OLV
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Optimal level of lung compliance during OLV | During the OLV phase of thoracic surgery
  A tidal volume (4-7 ml/kg PBW) where the pressure-volume loop reaches upper refection point and the peak airway pressure at or just below 30 cmH2O

SECONDARY OUTCOMES:
Postoperative pulmonary complication | 3 days after operation
  Composite endpoints of clinical diagnoses of pneumonia, bronchospasm, and/or ARDS), radiological diagnoses of atelectasis, pneumothorax, and/or pleural effusion, and therapies for respiratory insufficiency (need for prolonged therapy after end of surgery by providing supplemental oxygen, postoperative noninvasive ventilation, and/or reintubation with postoperative mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
1. Intraoperative ventilatory mechanic parameters
  2. Intraoperative hemodynamic measurements
  3. Intraoperative chest computer tomographic images
  4. Records of postoperative pulmonary complication rates